CLINICAL TRIAL: NCT02631889
Title: A Prospective, Randomized, Controlled Study to Assess the Effectiveness of Transcollation Technology to Reduce Bleeding in Lung Surgery
Brief Title: Study to Assess the Effectiveness of Transcollation Technology to Reduce Bleeding in Lung Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mohsen Ibrahim, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: V1/2015
Record Dates: First submitted 2015-12-10; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Blood Loss, Surgical
MeSH Terms: conditions — Blood Loss, Surgical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcollation technology (Experimental): the use of transcollation technology for hilium dissection during Lung surgery
  Interventions: Device: Transcollation technology
- Traditional Electrocautery (Active Comparator): The use of electrocautery for hilium dissection during lung surgery
  Interventions: Device: Traditional electrocautery

INTERVENTIONS:
Device: Transcollation technology — The use transcollation technology for dissection during lung surgery
  Arms: Transcollation technology
Device: Traditional electrocautery — The use of traditional Electrocautery for dissection during Lung Surgery
  Arms: Traditional Electrocautery

SUMMARY:
Major lung resection is one of the most common procedures performed in thoracic surgery, but it may involve considerable bleeding and the occasional need for a transfusion and/or reoperation for bleeding in specific cases. In addition, lysis of pleural-parenchymal adhesions and dissection can represent a challenge in patients who have undergone chemotherapy and/or radiation therapy, and in patients with bronchiectasis or COPD. Several intraoperative methods have been used to manage blood loss, including topical haemostatic agents, bipolar sealers or electrocautery. Transcollation technology (TT) consists of a disposable bipolar sealer that uses a radiofrequency coagulation system to deliver a saline solution that provides haemostatic sealing of soft tissue and bone and provides localized cooling without charring. Blood loss reduction has been previously described in several fields of surgery.

The primary end-point of the proposed trial is to assess if the ability of Transcollation Technology in reducing the proportion of patients showing bleeding perioperatively within the setting of a prospective randomized controlled trial.

The secondary end-point is to assess if Transcollation Technology is able to improve postoperative outcomes reducing the length of hospital stay.

DETAILED DESCRIPTION:
Study participation will start at signature of informed consent and each subject will be assessed preoperatively, within 4 weeks before surgery. A patient information leaflet will form the basis of discussions with the patient before written informed consent is obtained.

Patients will be evaluated intra-operatively, at 24 and 48 hours after surgery, and at discharge.

At the preoperative visit, the following information will be recorded on the patient's Case Report Form by a specialist Registrar:

* Patient number
* Patient initials
* Date of visit
* Demography (date of birth, sex, height, and weight)
* Preoperative FEV1 and % predicted FEV1
* Co-morbidities (chronic obstructive pulmonary disease [yes/no], current smoking habit [yes/no])
* levels of hemoglobin (preoperative, postoperative, 24 h, 48 h and discharged)
* perioperative complication.

Interventions

Patients undergoing Major Lung Surgery will be randomly assigned to one of two management strategies before the starting of the operation:

1. Electrocautery Using routine instrument for hilar dissection, hemostasis and lisys of eventual pleural adhesions.
2. Transcollation Technology Using Transcollation Technology for hilar dissection, hemostasis and lisys of eventual pleural adhesions.

Randomization Patients will be randomized in a 1:1 ratio to Transcollation technology (TT) or electrocautery. Patients will be allocated to the two different groups following a block randomization with sealed envelopes. This study is open-label: patients, investigators.

Allocation concealment The nature of the treatment precludes blinding of the surgeon administering the intervention. However, allocating, monitoring and measurement of all primary and secondary endpoints will be made by a dedicated investigator without the knowledge of, or reference to, the treatment allocation (electrocautery or Transcollation technology).

A dedicated investigator will provide a series of sealed envelopes, each containing a randomized treatment allocation. The operating surgeon will ascertain the treatment allocation for each eligible patient by opening the next available sealed randomization envelope. For each patient, the opened envelope will be attached to the Case Report Form for statistical analysis.

Sample Size Group sample sizes of 77 and 77 achieve 90% power to detect a difference of 65,0 ml of chest drain fluid at 24 h between the null hypothesis that both group means of chest drain fluid are 425,0 ml and the alternative hypothesis that the mean of group 2 is 360,0 ml with known group standard deviations of 124,0 ml, with a significance level (alpha) of 0,05 using a two-sided two-sample t-test. We consider a 10% of drop-out then we will recruit 170 patients.

ELIGIBILITY:
Inclusion Criteria:

* To be considered for enrollment, patients must:

  * be aged ≥ 18 years (of either gender)
  * have provided written informed consent prior to participation in the study
  * undergoing to major lung surgery with an open approach.

Exclusion Criteria:

* To be considered for enrollment, patients must not:

  * rethoracotomy
  * presence of pleural adhesions
  * coagulitive disorders or disease
  * have a known immune system disorder or immunodeficiency
  * be a participant in another interventional clinical trial or have received another investigational device or device within the last 30 days (donation of excised tissue [lung or parts of lymph nodes] for biological research may occur in the same patients)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Blood Loss, Milliliters (mL) | 24 hrs
  The mean quantity of chest drain fluids at 24 hours of patients in the Transcollation technology (TT) group compared with electrocautery group.

SECONDARY OUTCOMES:
Blood loss (g/dl) | 24 hrs
  hemoglobin level in the blood compared to the pre-operative level

OTHER OUTCOMES:
Length of hospital stay | 7 days
  Length of hospital stay (days), chest Drain duration and Heamoglobin variation of patients in the Transcollation technology (TT) group compared with electrocautery (EC) group.

CONTACTS AND LOCATIONS:
Overall Officials: Erino A Rendina, Professor, Study Chair — University of Roma La Sapienza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] S Hammond J, Muirhead W, Zaitoun AM, Cameron IC, Lobo DN. Comparison of liver parenchymal ablation and tissue necrosis in a cadaveric bovine model using the Harmonic Scalpel, the LigaSure, the Cavitron Ultrasonic Surgical Aspirator and the Aquamantys devices. HPB (Oxford). 2012 Dec;14(12):828-32. doi: 10.1111/j.1477-2574.2012.00547.x. Epub 2012 Aug 26. PMID 23134184
- [Background] Uchiyama A, Miyoshi K, Nakamura K. VIO soft-coagulation system for major pulmonary resections: results in 68 patients with primary lung cancer. Gen Thorac Cardiovasc Surg. 2011 Mar;59(3):175-8. doi: 10.1007/s11748-010-0709-5. Epub 2011 Mar 30. PMID 21448793
- [Background] Litle VR, Swanson SJ. Postoperative bleeding: coagulopathy, bleeding, hemothorax. Thorac Surg Clin. 2006 Aug;16(3):203-7, v. doi: 10.1016/j.thorsurg.2006.05.010. PMID 17004547
- [Background] Falez F, Meo A, Panegrossi G, Favetti F, La Cava F, Casella F. Blood loss reduction in cementless total hip replacement with fibrin spray or bipolar sealer: a randomised controlled trial on ninety five patients. Int Orthop. 2013 Jul;37(7):1213-7. doi: 10.1007/s00264-013-1903-8. Epub 2013 May 18. PMID 23685830